CLINICAL TRIAL: NCT03947281
Title: Almond Snacks and Satiety: a Randomized Intervention Trial Examining Acute and Chronic Effects
Brief Title: Snacks and Satiety
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: After delay due to pandemic, sponsor declined to continue funding.
Sponsor: USDA, Western Human Nutrition Research Center (U.S. Federal Agency)
Collaborators: Almond Board of California (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: FL107
Record Dates: First submitted 2019-05-09; First posted 2019-05-13 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Eating Behavior; Overweight; Obesity
Keywords: satiety; gastrointestinal hormones; appetite; Dietary fiber; food cravings
MeSH Terms: conditions — Feeding Behavior; Overweight; Obesity

STUDY DESIGN:
Intervention Model Description: The study will be a randomized, parallel design that includes an almond snack group and a cereal-based snack group. The intervention will be for 28 days. The almond intervention will be roasted almonds 56 grams/day. The cereal-based snack intervention will be the caloric equivalent.
Who Masked: Outcomes Assessor
Masking Description: Both the investigator and the participant will be aware of the group assignment. The persons handling the data and statistics will not be aware of the group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Almond snack (Experimental): The almond intervention will be roasted almonds 56 grams/day for 28 days. The caloric value is approximately 350 kcals.
  Interventions: Other: Almond snack
- Cereal-based snack (Experimental): The cereal-based intervention will be a mixture of dry cereal, pretzels, and bread sticks prepared by the Western Human Nutrition Research Center (WHNRC). The caloric value is approximately 350 kcals.
  Interventions: Other: Cereal-based snack

INTERVENTIONS:
Other: Almond snack — The almond intervention will be roasted, unsalted almonds provided at 56 g/day for 28 days. Almonds provide approximately 350 kcals/day.
  Arms: Almond snack
Other: Cereal-based snack — The cereal-based intervention will be a prepared mix of cereal, pretzels, and bread sticks prepared at the WHNRC. It will be provided at the level of 350 kcals per day for 28 days.
  Arms: Cereal-based snack

SUMMARY:
This study is designed to compare two types of snacks (almonds or a cereal-based snack), eaten between meals, on measures of appetite, including appetitive hormones, self-reported feelings of hunger and fullness, and food intake at a buffet meal or in the home environment. The investigators hypothesize that the acute responses of appetitive hormones to a meal challenge protocol will differ between almond and cereal-based snacks based on multivariate models of satiety that will be predictive of ad libitum food intake at a dinner meal as part of the meal challenge protocol. Further, the investigators will estimate if, under free-living conditions, self-selected and self-reported food intake will show appropriate energy compensation for the added calories of the snacks, and determine if one type of snack is superior to the other in this regard.

DETAILED DESCRIPTION:
This study will use a randomized, parallel design that includes an almond snack intervention and a cereal-based snack intervention group. The almond intervention will be roasted, unsalted almonds at a level of 56 grams per day for 4 weeks. The cereal-based intervention will be isocaloric snacks provided in the form of a mixture of dry cereal, pretzels, and bread sticks for 4 weeks. A satiety test protocol will be done at the beginning and the end of the intervention period. Each test day will include measures of satiety responses to two standard meals, two snacks (either almonds or cereal-based snacks), and a dinner buffet. The protocol to evaluate satiety signals include tonic measures that may signal homeostasis to the brain and evaluation of episodic signals that may drive food intake In addition, other modulators of satiety will be tested including evaluation of preferences for palatable foods, self-reports of cravings and satiety using questionnaires, and perceived hunger, fullness, desire to eat.

ELIGIBILITY:
Inclusion Criteria:

* Pre-menopausal
* Body Mass Index 25 - 39.9 kg/m2

Exclusion Criteria:

* Women who are post-menopausal or peri-menopausal
* BMI < 25 or > 40 kg/m2
* Allergies to tree nuts
* Using any hormonal contraception including oral contraceptive, contraceptive patch, contraceptive ring, contraceptive injection (e.g. Depo-Provera), or contraceptive implant (e.g. Nexplanon/Implanon)
* Menstrual cycle lengths < 25 days or > 45 days, or have amenorrhea, eumenorrhea, or polymenorrhea.
* Pregnant or nursing within the last 6 months, or plan to become pregnant during the trial
* Medical diagnoses of chronic diseases including cardiovascular or pulmonary diseases, renal disease, cancer, type 1 or type 2 diabetes mellitus, thyroid disease requiring medication, inflammatory bowel disease, irritable bowel disease, or those with recent major surgeries
* current medical diagnosis of polycystic ovarian syndrome (PCOS).

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2019-06-24 (Actual); Primary Completion 2022-08-08 (Actual); Study Completion 2022-08-08 (Actual)

PRIMARY OUTCOMES:
Baseline level and change in cholecystokinin | Baseline, 60 minutes before lunch meal, and 10, 30, 90, 150, 180, 210, 240, and 270 minutes after a lunch meal
  Cholecystokinin (CCK) measured in blood using an antibody based assay
Baseline level and change in peptide-YY | Baseline, 60 minutes before lunch meal, and 10, 30, 90, 150, 180, 210, 240, and 270 minutes after a lunch meal
  Peptide-YY (PYY) measured in blood using an antibody based assay
Baseline level and change in glucose-like peptide 1 | Baseline, 60 minutes before lunch meal, and 10, 30, 90, 150, 180, 210, 240, and 270 minutes after a lunch meal
  Glucose-like peptide 1 (GLP-1) measured in blood using an antibody based assay
Baseline level and change in gastric inhibitory peptide | Baseline, 60 minutes before lunch meal, and 10, 30, 90, 150, 180, 210, 240, and 270 minutes after a lunch meal
  Gastric inhibitory peptide (GIP) measured in blood using an antibody based assay
Baseline level and change in insulin | Baseline, 60 minutes before lunch meal, and 10, 30, 90, 150, 180, 210, 240, and 270 minutes after a lunch meal
  Insulin measured in blood using an antibody based assay
Baseline level and change in glucose | Baseline, 60 minutes before lunch meal, and 10, 30, 90, 150, 180, 210, 240, and 270 minutes after a lunch meal
  Glucose measured by standard chemistry in blood
Baseline level and change in oleoylethanolamide | Baseline, 60 minutes before lunch meal, and 10, 30, 90, 150, 180, 210, 240, and 270 minutes after a lunch meal
  Oleoylethanolamide measured by mass spectrometry in blood
Baseline level and change in ghrelin | Baseline, 60 minutes before lunch meal, and 10, 30, 90, 150, 180, 210, 240, and 270 minutes after a lunch meal
  Ghrelin measured in blood using an antibody based assay
Baseline level and change in leptin | Baseline, 60 minutes before lunch meal, and 10, 30, 90, 150, 180, 210, 240, and 270 minutes after a lunch meal
  Leptin measured in blood using an antibody based assay
Baseline level and change in orexin | Baseline, 60 minutes before lunch meal, and 10, 30, 90, 150, 180, 210, 240, and 270 minutes after a lunch meal
  Orexin measured in blood using an antibody based assay
Baseline level and change in endocannabinoid profiles | Baseline, 60 minutes before lunch meal, and 10, 30, and 150 minutes after a lunch meal
  Endocannabinoid profiles measured by mass spectrometry in blood
Baseline level and change in hunger | Baseline, every 30 minutes up to 480 minutes, and immediately before and after three meals
  Self-reported feelings of hunger measured on a visual analog scale. Responses will be a marked on an unsegmented line from 0 or "not at all" to 100 or "extremely."
Baseline level and change in satiety | Baseline, every 30 minutes up to 480 minutes, and immediately before and after three meals
  Self-reported feelings of fullness measured on a visual analog scale. Responses will be a marked on an unsegmented line from 0 or "not at all" to 100 or "extremely."
Change in food intake at a dinner meal | Week 1 and 4
  Calories consumed at a dinner meal following the satiety protocol

SECONDARY OUTCOMES:
Body composition reference measurement | Week 1
  Body composition (fat mass and fat-free mass in kg) will be measured once during the study using dual energy x-ray absorptiometry (DEXA)
Change in body weight | Weeks 0, 1, 2, 3, and 4
  measured in kg
Change in body fat | Weeks 0, 1, 2, 3, and 4
  measured in kg using multi frequency bioimpedance
Change in lean body mass | Weeks 0, 1, 2, 3, and 4
  measured in kg using multi frequency bioimpedance
Change in total body water | Weeks 0, 1, 2, 3, and 4
  measured in kg using multi frequency bioimpedance
Change in waist circumference | Week 0 and 4
  measured in cm
Change in hip circumference | Week 0 and 4
  measured in cm
Change in Food Choice | Baseline and following a lunch meal at Weeks 0 and 4
  Food choice computer-based tests from Leeds, United Kingdom, will be used to estimate explicit liking and implicit wanting for several different categories of foods.
Change in food craving | Week 0 and 4
  Food craving estimated from the questionnaire, Food Craving Inventory, on a 5 point likert scale
Change in self-reported satiety | Week 0 and 4
  Self reported satiety measured using the 5-factor satiety questionnaire. Scale is a generalized labeled magnitude scale of 150 mm Subscales include mental hunger, physical hunger, mental fullness, physical fullness, and satiation. Subscale scores will range from 0 to 150.
Power of food questionnaire | Week 0
  Power of food questionnaire measured once on a 5 point likert scale
Food addiction questionnaire | Week 0
  Yale food addiction questionnaire measured once on a 5-point likert scale
Eating behavior | Week 0
  Dutch eating behavior questionnaire measured once. Scale is a 5-point likert scale. Sub scales include restrained eating, emotional eating, and external eating. Scores will be reported separately for each subscale.
Three factor eating inventory | Week 0
  Three factor eating inventory questionnaire measured once. Instrument has three subscales, combining likert scales and true/false questions. Subscales include cognitive restraint (score can range from 0 to 21), disinhibition (score can range from 0 to 16) and hunger (score can range from 0 to 14).
Premenstrual Syndrome | Week 0
  Premenstrual Syndrome screening questionnaire measured once. Scale is a 4-point likert. Subscales for premenstrual syndrome (PMS) or premenstrual dysphoric disorder (PMDD), reported separately.
General health and well-being | Week 0
  The SF-36 General Health and Well-being questionnaire measured once
Usual physical activity | Week 0
  Physical activity estimated from the Stanford Brief Physical Activity questionnaire. Scale is categorical for two subscales: work physical activity and leisure time activity.
Change in metabolic rate | Baseline and 1 hour before lunch meal, 1 hour after lunch meal, and 1 hour after mid-afternoon snack
  Resting and post-prandial metabolic rate measured using indirect calorimetry.
Change in dietary intake | Ten dietary recalls collected at home during weeks 1-4
  Dietary intake estimated from 24-hour recall using a web based automated multi-pass method
Genetic risk of obesity | Week 1
  A polygenic risk score (PRS) indexing genetic predisposition to obesity using known obesity single nucleotide polymorphisms (SNPs).
Change in liver fat | Week 0 and 4
  Liver fat assessed from the Controlled Attenuation Parameter (CAP) computed from the liver stiffness measurement using the Fibroscan®
Change in liver stiffness | Week 0 and 4
  Liver stiffness assessed from the shear wave speed with pulse echo ultrasound using the Fibroscan®

CONTACTS AND LOCATIONS:
Locations (1):
- USDA, ARS, Western Human Nutrition Research Center, Davis, California, United States

IPD SHARING:
Plan to Share IPD: No